CLINICAL TRIAL: NCT05798858
Title: A Pilot Study for Implementation of First Trimester Screening of Aneuploidies in Campania Region
Acronym: PISTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Laura Sarno, Principal Investigator, Researcher, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 438/21
Record Dates: First submitted 2023-03-21; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Aneuploidy
Keywords: aneuploidy; screening; combined test; non invasive prenatal testing
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: NT+ NIPT (Active Comparator): Group A patients will undergo NT between 11+3 and 13+6 weeks. If the NT is <3.5 mm, the patient will be offered to continue the screening with NIPT.
  If NIPT comes back as positive result, the result will be confirmed by an invasive procedure (amniocentesis/villocentesis); if, on the other hand, the NIPT will give a negative result, the screening is concluded and the patient will not undergo further tests.
  Interventions: Diagnostic Test: NIPT
- Group B (Active Comparator): Combined test + NIPT (n=200) The patients of group A will undergo NT between 11+3 and 13+6 weeks, according to the same protocol foreseen for Group A.
  If the NT is <3.5 mm, the patient will be offered continuation of the screening using the combined test.
  In case of:
  High risk (1:2-1:100), the patient will be offered an invasive procedure (amniocentesis/villocentesis) Intermediate risk (1:101-1:1000), the patient will be offered NIPT, according to the protocol already described for Group A. In the event of a positive result, the patient will undergo an invasive procedure (amniocentesis/villocentesis ); in the case of negative NIPT, the screening is concluded and the patient will not undergo further tests.
  Low risk (>1:1000), screening ends and the patient will not undergo further tests.
  Interventions: Diagnostic Test: NIPT

INTERVENTIONS:
Diagnostic Test: NIPT — universal nipt in group a, NIPT for intermediate risk in Group B

SUMMARY:
The study aims to compare two different protocols for first trimester screening of aneuploidies, one based on nuchal translucency and NIPT and another one based on the integration between combined test and NIPT, in order to identify which is the most adequate for the Campania region.

In particular, a cost-benefit comparison will be made which will take into account for each method:

* Actual costs;
* Percentage of patients who agree to undergo the proposed screening and number of patients who undergo extra tests not included in the screening protocol;
* Post-invasive procedure miscarriage rate;
* False positives (fetuses undergoing an invasive procedure for a positive screen, which have a normal karyotype).

DETAILED DESCRIPTION:
INTRODUCTION Aneuploidies are pathologies characterized by an alteration in the number of chromosomes. They represent the most common form of fetal abnormalities.

The prenatal diagnosis of aneuploidy is currently based both on invasive diagnostic procedures (amniocentesis and CVS) and on non-invasive screening tests.

Invasive procedures are diagnostic tests, but they are burdened by quite high costs and by a risk of miscarriage, which is estimated at around 0.5-1%. For these reasons, these procedures can not offered to all pregnant patients.

The Bindi Decree in 1988 defined advanced maternal age (>35 years) as a sufficient indication to offer an invasive procedure. However, screening based on maternal age alone demonstrated very low sensitivity (about 35%) with a very high false positive rate (about 15%). Furthermore, if we consider the progressive increase in maternal age in the first pregnancy, we realize that the number of patients who fall into the high-risk group according to maternal age is extremely high. According to Cedap data 2013, around 25% of pregnant women were aged >35; this means that invasive procedures were offered to about 1 in 4 patients.

Over the years, aneuploidy screening has improved, first thanks to the introduction of biochemical markers (tri-tests and quadruple-tests) and, then, with the revolutionary advent of combined screening.

This screening is based on anamnestic data (maternal age, previous fetuses affected by aneuploidies), ultrasound data (measurement of nuchal translucency and fetal heart rate), biochemical data (dosage of free beta-hCG and PAPP-a: "DUO test" ) with a sensitivity of 90% and a false positive rate of about 4%.

Recently, cell free Dna testing has been introduce; this is a non-invasive test demonstrating high accuracy (99.7%) for Down syndrome and over 90% accuracy also for Trisomy 13 and 18. The main limitations of thus test are the high costs and the fact that without a good ultrasound screening, it does not allow the identification of severe fetal anomalies, easily detectable already in the first trimester of pregnancy (eg: anencephaly).

In 2017, the new Essential Levels of Assistance (LEA) have been approved subverting the now outdated Bindi Decree and introducing the combined test among the procedures that will be offered by the National Health System free of charge. Moreover, They underlined that access to invasive procedures should not based on maternal age alone, but on combined risk.

In Campania Region, a regional protocol for first trimester screening of aneuploidy has never been approved and patients can access both combined screening and cell free fetal DNA only in private settings.

Our project has as main objective the implementation of the screening for aneuploidies in Campania Region; moreover, we aim to compare two screening methods to define which one allows a better identification of the high-risk population to be destined for invasive procedures. In both cases, the nuchal translucency (NT) ultrasound is performed first, that is a service provided by the NHS; if this shows a value < 3.5 mm (99th percentile), one of the two possible procedures will be randomly offered:

* In one group, the fetal DNA test (NIPT) is carried out; if this is positive, an indication is given for the invasive test (villocentesis/amniocentesis).
* In the other, the combined test, financed by the research fund, is carried out first; if this highlights an intermediate risk, we proceed with NIPT, which if positive, directs us to amniocentesis.

MATERIAL AND METHODS Patients referred to the Mother & Child Department of theUniversity Hospital. Federico II of Naples to perform first trimester screenining ultrasound scan, will be included in the study.

Exclusion criteria: maternal age <18 years, lack of consent to participate in the study, twin pregnancy, ultrasound finding of a crown rump length >84 mm.

Patients will be recruited at the time of the first trimester screening ultrasound (nuchal translucency-NT), between 11+3 and 13+6 weeks of gestation.

If the patient decides to participate in the study, she will be asked to sign an informed consent. We will then proceed with the collection of all the anamnestic data necessary for the evaluation of the risk of aneuploidies which will be recorded in a dedicated database, in compliance with the privacy. In particular, the following information will be collected:

* Age of the patient;
* Previous fetuses affected by aneuploidy;
* Weight, height, ethnicity, presence of diabetes, type of conception (spontaneous, after the use of ovulation-inducing drugs, with intrauterine insemination, after homologous/heterologous medically assisted fertilization techniques).

All patients who decide to participate in the study will be counseled by a geneticist.

Patients will be randomized into two groups according to a 1:1 randomization scheme:

GROUP A: NT+ NIPT (n=200) Group A patients will undergo NT between 11+3 and 13+6 weeks. This scan will be performed by accredited operators according to the standards set by the Fetal Medicine Foundation (FMF) and by the Italian Society of Obstetrics and Gynecological Ultrasound (SIEOG).

The ultrasound examination is performed with transabdominal and/or transvaginal ultrasound, through the use of a real-time ultrasound equipped with a transabdominal and transvaginal transducer. During this examination, the following parameters will be evaluated, which will be used to calculate the combined risk:

* Crown rump length (CRL): this measurement is obtained from a sagittal scan of the fetus, which must assume a neutral position, with the head in line with the column (not hyperflexed or hyperextended). CRL measurement is used to redate pregnancy according to ultrasound gestational age; this re-dating is not carried out for pregnancies obtained after medically assisted fertilization in which the dating of the pregnancy is certain. NT ultrasound can only be performed for CRLs between 45 and 84 mm. In the case of CRL <45 mm, a new appointment will be scheduled for the patient, while, in the case of CRL >84 mm, the patient will be excluded from the study.
* Fetal heart rate (FHR), obtained from a cross-sectional scan of the fetus at the level of the tricuspid valve.
* Nuchal translucency (NT): the measurement of NT is obtained in sagittal scan of the fetus which must appear horizontally on the screen, with obtaining the image of the fetal profile (reference points: visualization of the nose, the palate must have a rectangular shape and the frontal process of the maxilla should not be visualised, visualization of the diencephalon). Ideal images should include only the fetal head and upper chest. The magnification of the image must be such that each movement of the caliper produces a change in the measurement of 0.1 mm. Measurements should be taken with the inner edge of the horizontal line of the calipers positioned on the line defining the thickness of the nuchal translucency. The horizontal bar of the calipers should not protrude into the anechoic space of the nuchal translucency. It is necessary to distinguish the fetal skin from the amnion.

Minor ultrasound markers (nasal bone, ductus venosus, tricuspid regurgitation) will not be included in the combined risk.

All ultrasound data and images will be saved in a special program dedicated to ultrasound storage and reporting.

If the NT is >3.5 mm (99th centile), the patient will be offered an invasive procedure (amniocentesis or CVS).

If, on the other hand, the NT is <3.5 mm, the patient will be offered to continue the screening with NIPT.

A dedicated midwife will complete a specific request and collect a blood sample that will be sent to the laboratory.

If NIPT comes back as positive result, the result will be confirmed by an invasive procedure (amniocentesis/villocentesis); if, on the other hand, the NIPT will give a negative result, the screening is concluded and the patient will not undergo further tests.

GROUP B: Combined test + NIPT (n=200) The patients of group A will undergo NT between 11+3 and 13+6 weeks, according to the same protocol foreseen for Group A.

If the NT is >3.5 mm (99th centile), the patient will be offered an invasive procedure (amniocentesis or CVS).

If the NT is <3.5 mm, the patient will be offered continuation of the screening using the combined test.

The execution of this test involves the compilation of a special form by a dedicated midwife, who will also take a blood sample from the patient. The sample will be send to the DAI of Laboratory and Transfusion Medicine of the AOU Federico II.

The test involves the dosing of two placental products, free beta-hCG and PAPP-a, which will be carried out through the use of accredited equipment, already available at the DAI of Laboratory and Transfusion Medicine of AOU Federico II . The patient will be notified of a risk calculated according to the algorithm proposed by the FMF, which brings together the patient's basic risk (maternal age, previous affected fetus), ultrasound data (NT, CRL, FHR) and the two biochemical markers (free beta -hCG and PAPP-a).

In case of:

* High risk (1:2-1:100), the patient will be offered an invasive procedure (amniocentesis/villocentesis)
* Intermediate risk (1:101-1:1000), the patient will be offered NIPT, according to the protocol already described for Group A. In the event of a positive result, the patient will undergo an invasive procedure (amniocentesis/villocentesis ); in the case of negative NIPT, the screening is concluded and the patient will not undergo further tests.
* Low risk (>1:1000), screening ends and the patient will not undergo further tests.

Outcome collection The collected data will include the outcome of the pregnancy (spontaneous abortion, voluntary termination of pregnancy, intrauterine fetal death, live birth) and the cases of aneuploidies found (by karyotype in patients undergoing amniocentesis or CVS or direct postnatal assessment if prenatal karyotype is not known). All those that occur within seven days following the procedure will be considered post-procedure abortions.

STATISTIC ANALYSIS The statistical analysis will be conducted through the SPSS 27.0 statistical analysis program (Chicago Inc.) All data relating to descriptive analysis will be reported as median (interquartile range-IQR) for continuous variables, and absolute frequency (percentage) for categorical variables.

The comparison between continuous variables will be performed through the parametric test T-Student and the non-parametric test of Mann-Whitney. The comparison between categorical variables will make use of the Chi-squared test and Fisher's exact test.

Correlations between parameters will be evaluated through the Pearson correlation coefficient.

ETHICAL CONSIDERATIONS The study has been approved by local ethical committee (IRB 438/21)

EXPECTED RESULTS AND IMPACT We expect this study to clarify which method is more feasible in terms of diagnostic accuracy and costs, in order to provide the basis for the identification of a screening method to be implemented in Campania Region.

ELIGIBILITY:
Inclusion Criteria:

* all patients referred to our hospital for first trimester screening scan

Exclusion Criteria:

* maternal age<18
* twin pregnancies
* lack of a signed consent form

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
compliance to the screening | up to 9 months
  percentage of patients not performing test not included in arm protocol

SECONDARY OUTCOMES:
spontaneous abortions | up to seven days
  percentage of post-procedure spontaneous abortions
sensitivity and specificity of two protocols | up to 9 months
  sensitivity and specificity of two protocols
total costs | up to 3 months
  cost- effective analysis of two protocols

CONTACTS AND LOCATIONS:
Locations (1):
- University Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No